CLINICAL TRIAL: NCT03281278
Title: A Prospective Study of Application of Platelet Mapping in HBV-related Acute-on-chronic-liver Failure in China
Status: Completed | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 003
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2018-04

CONDITIONS: Thrombelastography,Acute on Chronic Liver Failure, Platelet
Keywords: Thrombelastography,acute on chronic liver failure, platelet
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: standard treatment — standard medical treatment

SUMMARY:
Ineffective hemostasis or a paradoxical prothrombotic state of Acute-on-chronic liver disease (ACLF) has been well established. Thrombelastography measures the dynamics of thrombin production and provides a global assessment of coagulation incorporating the cumulative effect of the interactions at various levels between plasma components and cellular component of coagulation. And through the platelet mapping, it can help provide a picture of patients' function of platelet. This study aims to explore the predictive role of platelet mapping in ACLF prognosis, organ failure developments and short term mortality.

ELIGIBILITY:
Inclusion Criteria:

* patient with previously diagnosed or undiagnosed HBV related chronic liver disease/cirrhosis
* INR≥1.5 and total bilirubin≥85μmol/L

Exclusion Criteria:

* INR≤1.5 or total bilirubin≤85μmol/L;
* underlying chronic liver disease was other than chronic HBV infection related;
* those who had hepatocellular carcinoma or other types of malignancies;
* obstructive biliary diseases or other disease lead to bilirubin evaluation;
* those who had acute hemorrhage one week before admission
* those who received platelet, cryo transfusion or plasmapheresis one week before admission
* using steroid or immunosuppressant or antiplatelet or anticoagulant drugs in 4 weeks
* any kind of decompensation which persisted over a month
* pregnancy and breastfeeding
* those who received liver transplantation or kidney transplantation;
* combine with other disease lead to organ failure including heart failure (NYHA IV),respiratory failure（PaO2<60mmHg),renal insufficiency(CKD 5) and conscious disturbance (GCS<8)
* readmission;
* death within 24 hours.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HBV-related chronic liver disease, International Normalized Ratio (INR)≥1.5 and total bilirubin≥85μmol/L
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2018-08-13 (Actual)

PRIMARY OUTCOMES:
28-day mortality | 28-day
  death within 28-day

SECONDARY OUTCOMES:
28-day progression | 28-day
  progressed to EASL defined ACLF
90-day mortality | 90-day
  death within 90-day

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China